CLINICAL TRIAL: NCT05975658
Title: WIReD: Wireless Interstage Remote Device Study
Acronym: WIReD
Status: Completed | Type: Observational
Sponsor: Children's Mercy Hospital Kansas City (Other)
Collaborators: Gabi SmartCare (Industry)
Responsible Party: Principal Investigator, Lori Erickson, Director, Remote Health Solutions, Children's Mercy Hospital Kansas City
Other Study IDs: STUDY00002554
Record Dates: First submitted 2023-07-27; First posted 2023-08-04 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Congenital Heart Disease in Children; Vital Signs; Pediatrics; Remote Monitoring
Keywords: Pediatric; Physiologic vital signs

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: Gabi SmartCare Pediarity System [Gabi Band, Gabi Monitor App, Gabi Analytics] — Gabi SmartCare has created a monitoring system named Pediarity System that obtains pediatric vitals data through non-invasive means through a Gabi band. When paired with a proprietary algorithm and software - Gabi Analytics - the cloud-based platform measures blood oxygen levels, pulse rate (and variability), respiratory rate, actigraphy, inter-beat interval, and tracking for the time the device is worn (or not worn by the child). Three LEDs on the monitor are used for capturing this information. Peak wavelengths for the red, infrared, and green LEDs operate at 660nm, 950nm, and 526nm respectively. The Gabi band features an optical front end coupled with an analog front end using 24 bits. Bluetooth data transmission is utilized on a mobile phone application with a tablet-based system in a CSV format for the purpose of offline data processing.

SUMMARY:
A mixed-methods study will be used to evaluate the use of standard of care periodic pulse oximetry by parents/LAR and the feasibility of the collection of physiologic data related to the use of the Pediarity System. This system includes the Gabi Band and software platform (Gabi Analytics).

DETAILED DESCRIPTION:
After enrollment, parents will be taught by the study team on the use of the Pediarity System which includes the placement of the Gabi Band and the use of the Gabi Wi-Fi monitor application for data transfer. This education by the study team will ensure uniform training and preliminary understanding with teach back on the use of the Gabi band and Gabi Wi-Fi monitoring application. Parents can ask the study team any use and/or technical questions during this time period. All clinical care questions from standard of care monitoring will go to the CHAMP healthcare team. If parents/LARs have a clinical concern from a value on the Pediarity System - they will be referred to use their standard of care pulse oximetry before any clinical intervention and care is recommended by the healthcare team. The study team will not make any healthcare or diagnostic recommendations during the monitoring period based on any Pediarity System data.

The study team will educate parents and LARs on the Pediarity System. This system does not replace any use of their standard of care pulse oximetry and CHAMP videos. Parents may place the Gabi band on their child and use the Pediarity System at any frequency they choose in the home setting for a length of approximately one month at home (to coordinate when they return to the study site for a care visit). Parents can email or Teams call the study team directly (during daytime hours M-F) for any technical questions during this the study period. The study team will evaluate clinical data only at the conclusion of the study period and qualitative feedback from the parents will be gathered.

ELIGIBILITY:
Inclusion Criteria:

* Study participants will be parent-child dyads - pediatric patients who have been diagnosed with congenital, arrhythmic, or acquired heart disease at Children's Mercy Kansas City.
* Age criteria for children: after birth and who are less than two years of age at the time of being approached.
* The child of the parent-child dyad must be planned from the clinical standpoint prior to approach for discharge home with standard of care oxygen saturation/heart rate/pulse oximeter for remote patient monitoring population - and followed with the CHAMP application in the home setting.
* CHAMP App CM IRB 15030113 - Pediatric patients may be followed by the CHAMP Clinical team or enrolled in the CHAMP App Cardiac Study

Exclusion Criteria:

* Over two years of age at the time of being approached for study participation.
* Families that do not speak English or Spanish (languages supported by the devices).
* Families that do not have access to a Wi-Fi network at home.

Max Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Maximum of 15 infants in the congenital, arrhythmic, or acquired heart disease population to be enrolled at Children's Mercy Hospital Kansas City.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2023-09-30 (Actual); Primary Completion 2024-12-03 (Actual); Study Completion 2024-12-03 (Actual)

PRIMARY OUTCOMES:
Parental Experience Evaluation | 3-6 Weeks
  Rigorously explore the parental experience of utilizing a continuous pediatric wireless device for monitoring at home pulse oximetry compared with standard of care periodic pulse oximetry through parent interviews.

SECONDARY OUTCOMES:
Data Transfer Rate Evaluation | 3-6 Weeks
  Evaluate the rate of data transfer from a wireless continuous monitoring device night ± daytime vs. standard of care periodic pulse oximetry.
Stakeholder Experience Assessment | 3-6 Weeks
  Assess the technology experience for stakeholders with a wireless continuous monitoring device at home vs. standard of care periodic pulse oximetry using healthcare provider interviews to discuss outcome experience.
Data Threshold Event Rate Evaluation | 3-6 Weeks
  Evaluate the rate of data threshold events with continuous remote device monitoring at home vs. intermittent pulse oximetry via standard of care periodic pulse oximetry.
Satisfaction with the System | 3-6 weeks
  Using the System Usability Survey (SUS) Strongly Disagree to Strongly Agree 1-7
Effectiveness with the System | 3-6 weeks
  Using the System Usability Survey (SUS) Strongly Disagree to Strongly Agree 1-7
Comfort with the System | 3-6 weeks
  Using the System Usability Survey (SUS) Strongly Disagree to Strongly Agree 1-7
Easy to use the System | 3-6 weeks
  Using the System Usability Survey (SUS) Strongly Disagree to Strongly Agree 1-7
Easy to find information within the System | 3-6 weeks
  Using the System Usability Survey (SUS) Strongly Disagree to Strongly Agree 1-7
Visualization of information within the System | 3-6 weeks
  Using the System Usability Survey (SUS) Strongly Disagree to Strongly Agree 1-7
Clear organization of information within the System | 3-6 weeks
  Using the System Usability Survey (SUS) Strongly Disagree to Strongly Agree 1-7
Functions of the System | 3-6 weeks
  Using the System Usability Survey (SUS) Strongly Disagree to Strongly Agree 1-7

CONTACTS AND LOCATIONS:
Overall Officials: Lori Erickson, PhD, Principal Investigator — Director, Remote Health Solutions Children's Mercy
Locations (1):
- Children's Mercy Hospital, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Gabi SmartCare Website — https://gabismartcare.com/